CLINICAL TRIAL: NCT05664477
Title: PhytoSERM Efficacy to Prevent Menopause Associated Decline in Brain Metabolism and Cognition: A Double-Blind, Randomized, Placebo-Controlled Phase 2 Clinical Trial
Brief Title: PhytoSERM to Prevent Menopause Associated Decline in Brain Metabolism and Cognition
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Roberta Brinton (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Cornell University (Other); ADM Diagnostics (Unknown)
Responsible Party: Sponsor-Investigator, Roberta Brinton, Regents Professor and Director of the Center for Innovation in Brain Science, University of Arizona
Organization: University of Arizona (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Phyto-2022-01; R01AG075122 (NIH)
Record Dates: First submitted 2022-09-08; First posted 2022-12-23 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Menopause; Cognitive Change; Brain Disorder, Metabolic
MeSH Terms: conditions — Brain Diseases, Metabolic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PhytoSERM group (Experimental): PhytoSERM 50mg tablet composed of the phytoestrogens daidzein, genistein and S-equol, administered orally every day for 24 weeks.
  Interventions: Dietary Supplement: PhytoSERM
- Placebo group (Placebo Comparator): Placebo product with identical shape, size and color with absence of daidzein, genistein, and S-equol. Administered orally every day for 24 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Dietary Supplement: PhytoSERM — PhytoSERM is a dietary supplement containing equal amounts of genistein (16.7 mg ± 10%), daidzein (16.7 mg ± 10%) and S-equol (16.7 mg ± 10%).
  Arms: PhytoSERM group
Drug: Placebo — Placebo product with identical shape, size and color will be produced with absence of S-equol, daidzein and genistein. Ingredients include calcium carbonate, comprecel M102, croscarmellose sodium, stearic acid, Zeofree 5162, magnesium stearate, carnauba wax, coating cellulose clear (PEG), coating white (PEG), water.
  Arms: Placebo group

SUMMARY:
This is a proof-of-concept phase 2 clinical trial to investigate the safety and effect of the phytoestrogenic supplement PhytoSERM on regional brain metabolism by fluorine-18 fluorodeoxyglucose positron emission tomography (18F-FDG-PET) in peri- and postmenopausal women. The investigators hypothesize that there will be a significant difference between the PhytoSERM group and placebo group in glucose brain metabolism.

DETAILED DESCRIPTION:
This is a double-blinded, randomized, placebo-controlled, parallel designed, proof-of-concept phase 2 clinical trial to determine effect of PhytoSERM in regional brain metabolism, cognition and vasomotor symptoms in menopausal women. PhytoSERM or placebo pills will be administered orally once a week over 24 weeks. Safety and tolerability will also be assessed over the duration of the study.

To determine eligibility, all participants will undergo cognitive assessment, physical and neurological examination, imaging scans, electrocardiogram (ECG), clinical/safety laboratory assessment, and interviews. After a 2-4-week screening period, participants will be randomized to study intervention (PhytoSERM 50mg administered orally, once per day) or matching placebo, in a 1:1 allocation. Brain imaging to evaluate the primary endpoint (standardized uptake value ratio (SUVR) by FDG-PET) will be conducted at screening and 24 weeks (6 months). Study participants will be asked to complete a total of 7 study visits. All participants will be enrolled at a single site, at the Alzheimer's Prevention Program (APP) at Weill Cornell Medical Centre (WCMC, New York).

This study protocol will include an embedded single-dose, 24-hour pharmacokinetic (PK) study in a subset of 12 participants which will begin after the first dose of the study intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Peri- or postmenopausal women with the latter defined as last menstrual period (LMP) completed ≥ 60 days and ≤ 4 years, per the Stages of Reproductive Aging Workshop (STRAW) criteria.
2. Age 45-60 years.
3. Presence of hot flashes ≥ 7 per day.
4. In good general health as evidenced by medical history.
5. Clinical laboratory values must be within normal limits or, if abnormal, must be judged to be not clinically significant by the investigator.
6. No medical contraindications to study participation.
7. Stable medications for 4 weeks prior to the baseline visits.
8. Provision of signed and dated informed consent form.
9. Stated willingness to comply with all study procedures and availability for the duration of the study.
10. Ability to take oral medication and be willing to adhere to the PhytoSERM regimen.
11. For females of reproductive potential: Negative pregnancy test and use of highly effective contraception by male partner for at least 1 month prior to screening and agreement to use such a method during study participation.
12. Fluent in English or Spanish.

Exclusion Criteria:

1. Known allergies to isoflavones or soy-based products.
2. Evidence of cognitive impairment on the Mini-Mental State Examination (total score < 27).
3. Pregnancy
4. Use of estrogen or progestin compounds within 8 weeks of baseline.
5. Use of investigational agent within 12 weeks of baseline.
6. Concurrent neurologic, systemic, or psychiatric disease that would influence cognition or ability to provide informed consent and to participate.
7. Known or suspected estrogen-dependent neoplasia, active neoplastic disease, history of breast cancer, or at risk of developing breast cancer, endometrial hyperplasia.
8. History of epilepsy, focal brain lesion, head injury with loss of consciousness or Diagnostic and Statistical Manual of Mental Disorders (DSM IV) criteria for any major psychiatric disorder including psychosis, major depression, bipolar disorder, alcohol or substance abuse.
9. Thrombophlebitis, thrombosis, thromboembolic disorders, myocardial infarction, ischemic heart disease, cerebrovascular accident, stroke, transient ischemic attack (TIA).
10. Current use of tobacco or a history of alcohol abuse.
11. Use of drugs, herbs, or dietary supplements to treat menopausal or cognitive symptoms less than 8 weeks prior to baseline.
12. Evidence of any significant clinical disorder or laboratory finding.
13. Known allergy to soy-derived products/ proteins or branded over the counter products; hypersensitivity to estrogens or progestins.
14. Visual and auditory acuity inadequate for neuropsychological testing
15. Inability to undergo MRI scans
16. Inability to undergo PET scans

Ages: 45 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-01-10 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Standardized uptake value ratio (SUVR) by 18F-FDG PET | Baseline to 24 weeks
  Regional brain glucose metabolism SUVR

SECONDARY OUTCOMES:
Trail Making Test (TMT) | Baseline to 24 weeks
  The TMT is scored by how long it takes to complete the test. For TMT-B, an average score is 75 seconds, and a deficient score is greater than 273 seconds. Less is better.
List Sorting Working Memory Test | Baseline to 24 weeks
  Test scores consisted of combined total items correct on the one- and two-list versions of the task (maximum 28). The raw sum score is then transformed to a standardized t-metric. More is better.
Picture Sequence Memory Test | Baseline to 24 weeks
  Maximum raw score of 48 for ages 20-60 years. More is better.
Auditory Verbal Learning Test | Baseline to 24 weeks
  The Rey is scored by taking the sum of the number of words recalled across all trials (possible range is 0-45 words).
Oral Symbol Digit Test | Baseline to 24 weeks
  The Oral Symbol Digit Test is scored as the number of items answered correctly in 120 seconds (possible range is 0-144).
Hot flash Frequency Composite | Baseline to 24 weeks
  Hot flash frequency and severity scores. Less is better.
Menopause Rating Scale (MRS) Score | Baseline to 24 weeks
  The total score of the MRS ranges between 0 (asymptomatic) and 44 (highest degree of complaints).
Pittsburgh Sleep Quality Index | Baseline to 24 weeks
  A global sum of "5" or greater indicates a "poor" sleeper.
Positive and Negative Affect Scale | Baseline to 24 weeks
  Positive and negative affect items are summed separately and range from 0 to 50 with higher scores indicating higher positive affect and higher negative affect respectively.
Beck Depression Inventory - II | Baseline to 24 weeks
  Maximum score is 63. Higher scores represent greater depressive symptoms.
Pharmacokinetics: Peak Plasma Concentration (Cmax) | Baseline
  The highest concentration of each phytoestrogen in the blood after a dose is given.
Pharmacokinetics: Time of peak concentration (tmax) | Baseline
  Time required to achieve peak plasma levels.
Pharmacokinetics: Half-life (t1/2) | Baseline
  The time required for plasma concentration of phytoSERMs to decrease by 50%
Pharmacokinetics: Area under the plasma concentration versus time curve (AUC) | Baseline
  The concentration of phytoSERMs in blood plasma as a function of time. Gives insight into the extent of exposure to phytoSERM and its clearance rate from the body.

OTHER OUTCOMES:
Regional brain volume | Baseline to 24 weeks
  T1-weighted volumetric MRI (mm3).
Fractional Anisotropy | Baseline to 24 weeks
  Multi-band multi-shell Diffusion Tensor Imaging (DTI) to measure changes in white matter tract integrity.
Quantitative anisotropy | Baseline to 24 weeks
  DTI to measure changes in white matter tract integrity. The amount of anisotropic spins that diffuse along the fiber orientation.
Functional connectivity | Baseline to 24 weeks
  Resting state functional MRI (rs-fMRI) to measure changes in intrinsic connectivity, which also correlates to neuronal function.
Cerebral blood perfusion | Baseline to 24 weeks
  Arterial spin labeling (ASL) to measure changes in cerebral blood flow, which correlates to neuronal function.
Inflammatory Biomarker: Cytokines | Baseline to 24 weeks
  Change in laboratory value in inflammatory cytokines (Interleukin-6)
Lipid biomarker: Total Cholesterol | Baseline to 24 weeks
  Laboratory value of total cholesterol in blood
Plasma Glucose | Baseline to 24 weeks
  Laboratory value of glucose in plasma
Diabetic biomarker: Hemoglobin A1C (HbA1c) | Baseline to 24 weeks
  Laboratory value
Menopause biomarker: Estradiol | Baseline to 24 weeks
  Laboratory values
Menopause biomarker: Follicle-Stimulating Hormone (FSH) | Baseline to 24 weeks
  Laboratory values

CONTACTS AND LOCATIONS:
Overall Officials: Roberta D Brinton, PhD, Principal Investigator — University of Arizona; Gerson D Hernandez, MD, MPH, Principal Investigator — University of Arizona
Locations (1):
- The Alzheimer's Prevention Program / Weill Cornell Medicine, New York, New York, United States

REFERENCES:
- [Background] Hernandez G, Zhao L, Franke AA, Chen YL, Mack WJ, Brinton RD, Schneider LS. Pharmacokinetics and safety profile of single-dose administration of an estrogen receptor beta-selective phytoestrogenic (phytoSERM) formulation in perimenopausal and postmenopausal women. Menopause. 2018 Feb;25(2):191-196. doi: 10.1097/GME.0000000000000984. PMID 28926513
- [Background] Schneider LS, Hernandez G, Zhao L, Franke AA, Chen YL, Pawluczyk S, Mack WJ, Brinton RD. Safety and feasibility of estrogen receptor-beta targeted phytoSERM formulation for menopausal symptoms: phase 1b/2a randomized clinical trial. Menopause. 2019 Aug;26(8):874-884. doi: 10.1097/GME.0000000000001325. PMID 30889096